CLINICAL TRIAL: NCT01420263
Title: Re-feeding Residuals Versus Feeding Fresh Formula/Milk for Feeding Intolerance in Premature Infants
Brief Title: Re-feeding Gastric Residuals in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ariel Salas, MD, Fellow Instructor, Department of Pediatrics, Division of Neonatology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAB Neo 004
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Premature; Infant, Light-for-dates
Keywords: premature infant; feeding; residuals; fresh feeds; full feeds; digestive system
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Re-feeding gastric residuals (Active Comparator): In the presence of significant gastric residuals (more than 1/3 of previous feed or > 2ml), residual volumes will be re-fed if the physician decision is to continue feeds as scheduled in the absence of other clinical signs and symptoms of feeding intolerance. This practice will be continued until full enteral feeding is achieved and maintained for a minimum of 48 hours.
  Interventions: Procedure: Re-feeding residuals
- Fresh feeding breastmilk/formula only (Active Comparator): In the presence of significant gastric residuals (more than 1/3 of previous feed or > 2ml), residual volumes will be discarded and fresh breast milk or formula will be fed if the physician decision is to continue feeds as scheduled in the absence of other clinical signs and symptoms of feeding intolerance. This practice will be continued until full enteral feeding is achieved and maintained for a minimum of 48 hours.
  Interventions: Procedure: Fresh Feeding Breastmilk or Formula only

INTERVENTIONS:
Procedure: Re-feeding residuals — In the presence of significant gastric residuals (more than 1/3 of previous feed or > 2ml), residual volumes will be re-fed if the physician decision is to continue feeds as scheduled in the absence of other clinical signs and symptoms of feeding intolerance. This practice will be continued until full enteral feeding is achieved and maintained for a minimum of 48 hours.
  Arms: Re-feeding gastric residuals
Procedure: Fresh Feeding Breastmilk or Formula only — In the presence of significant gastric residuals (more than 1/3 of previous feed or > 2ml), residual volumes will be discarded and fresh breastmilk or formula will be fed if the physician decision is to continue feeds as scheduled in the absence of other clinical signs and symptoms of feeding intolerance. This practice will be continued until full enteral feeding is achieved and maintained for a minimum of 48 hours.
  Arms: Fresh feeding breastmilk/formula only

SUMMARY:
The purpose of this study is to determine whether re-feeding of gastric residuals reduces the time needed to establish full enteral feedings in premature infants. Infants with gestational ages 23-28 weeks at birth will be randomized within one week to receive either gastric residuals or fresh formula or breastmilk whenever significant residuals during feeding advancement require clinical assessment for continuing feedings. Primary outcome measure is time to establish full enteral feedings (120cc/kg/day).

DETAILED DESCRIPTION:
Infants with gestational ages 23-28 weeks at birth will be randomized within one week to receive either gastric residuals or fresh formula or breastmilk whenever significant residuals during feeding advancement require clinical assessment for continuing feedings. Feeding advancement determined by clinical physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age between 23.0 and 28.6 weeks;
2. Receiving intravenous fluids but not enteral nutrition more than trophic feeds;
3. Written informed consent from the parents

Exclusion Criteria:

1. Major congenital/chromosomal anomalies;
2. Moribund infant with low likelihood of survival, in the opinion of the clinical team

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Time to establish full enteral feeding | Birth to 28 days
  Time required to reach enteral feeding at 120cc/kg/day

SECONDARY OUTCOMES:
Feeding intolerance | Birth to 28 days
  Feeding intolerance defined as interruption or cessation of enteral feeds for a perod greater than 12 hours for presence of bloody gastric residuals or an abnormal abdominal examination.
Episodes of feeding intolerance resulting in a interruption or cessation of progression of enteral feeds for a period of < 12 hours. | Birth to 28 days
  Number of episodes of feeding intolerance resulting in an interruption or cessation of progression of enteral feedings for a period of < 12 hours.
Number of days receiving parenteral nutrition | Birth to 28 days
  Total number of days or partial day receiving parenteral nutrition
Duration of hospital stay | Birth to 120 days or discharge, whichever occurs first.
  Length of hospital stay in days
Diagnosis of necrotizing enterocolitis | Birth to 120 days or discharge, whichever occurs first.
  Diagnosis of necrotizing enterocolitis, Bell's Staging II-IV
Diagnosis of intestinal perforation | Birth to 120 days or discharge, whichever occurs first
  Diagnosis of intestinal perforation between birth and 120 days or discharge, whichever occurs first.
Death | Birth to 120 days
  Death prior to 121 days of age.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel A Salas, MD, Principal Investigator — University of Alabama at Birmingham; Namasivayam Ambalavanan, MD, Study Director — University of Alabama at Birmingham; Waldemar A Carlo, MD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Salas AA, Cuna A, Bhat R, McGwin G Jr, Carlo WA, Ambalavanan N. A randomised trial of re-feeding gastric residuals in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2015 May;100(3):F224-8. doi: 10.1136/archdischild-2014-307067. Epub 2014 Dec 31. PMID 25552280